CLINICAL TRIAL: NCT05726773
Title: The Effect of Robot Assisted Hand Therapy on Hand Functions and Quality of Life in Patients With Spinal Cord Injury: A Randomized Controlled Study
Brief Title: The Effect of Robot Assisted Hand Therapy in Patients With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, assistant professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SATETRA
Record Dates: First submitted 2023-01-31; First posted 2023-02-14 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Tetraplegia
Keywords: Tetraplegia; Spinal cord injury; Robotic assisted therapy; Hand rehabilitation
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot Assisted Therapy Group (Experimental): In the RAT group, it was planned to perform robotic rehabilitation with a hand-finger robot [Amadeo (Tyromotion, Graz, Austria)] for 30 minutes for both upper extremities, accompanied by a physiotherapist who is trained in robotic rehabilitation and has at least 5 years of experience. In robotic rehabilitation, continuous passive range of motion (CPM), active assistive exercises and assistive continuous passive range of motion (CPM Plus) programs will be used.
  Interventions: Procedure: Robot Assisted Therapy; Procedure: Conventional Therapy
- Conventional Therapy Group (Active Comparator): In the Conventional Therapy group, an exercise program consisting of passive and active assistive range of motion exercises, strengthening exercises and task-oriented exercises for 30 minutes for both hands was planned, accompanied by a physiotherapist experienced in spinal cord injury rehabilitation for at least 5 years.
  Interventions: Procedure: Conventional Therapy

INTERVENTIONS:
Procedure: Robot Assisted Therapy — In robotic rehabilitation, continuous passive range of motion (CPM), active assistive exercises and assistive continuous passive range of motion (CPM Plus) programs will be used.
  Arms: Robot Assisted Therapy Group
Procedure: Conventional Therapy — In the Conventional Therapy group, an exercise program consisting of passive and active assistive range of motion exercises, strengthening exercises and task-oriented exercises for 30 minutes for both hands was planned, accompanied by a physiotherapist experienced in spinal cord injury rehabilitation for at least 5 years.

SUMMARY:
Considering the scarcity of studies on robotic hand therapy, it has been seen that larger-scale and long-term follow-up studies are needed. In this study, our aim is to compare the effects of robot-assisted hand therapy and conventional physiotherapy on hand functions and quality of life in patients with spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is considered one of the most devastating injuries that cause lifelong disability.Among the impaired functions, upper extremity function is one of the most important goals of rehabilitation for these individuals.Hand functions are among the most important determinants of independence.Some studies have reported that in more than half of people with tetraplegia, restoring arm and hand function will improve quality of life.Therefore, small improvements in upper extremity function can make a clinically significant difference in feeding, bathing, transferring and other functional activities.Given that the majority of individuals with spinal cord injuries are in their most productive years and life expectancy approaches that of the healthy population, more aggressive treatment strategies that focus on improving peripheral muscle control and recovery of the central nervous system (CNS) are needed.Recently, treatment based on the 'motor learning theory' has been reported to be effective in the recovery of impaired upper extremity function.It has been shown that by repetitive movements as intense as possible to help achieve the ultimate goal of optimum movement, patients are able to learn motor skills that lead to CNS recovery.It has also been suggested that repetitive and activity-based exercise may facilitate recovery after spinal cord injury by inducing practice-dependent brain and spinal cord plasticity.Therefore, repetitive, intensive, and activity-based upper extremity rehabilitative therapy can help improve impaired upper extremity function.In this context, robotic therapy (RT) may be an alternative way of delivering rehabilitative therapy to patients with tetraplegia, as RT can deliver consistently high-intensity, high-repetition, and task-specific training with less effort compared to conventional therapy.

ELIGIBILITY:
Inclusion criteria:

* Mini mental test score >15
* Able to understand the commands
* Had a function between 1 and 4 in at least one of the key muscle strengths in at least one hand.

Exclusion Criteria:

* Patients with persistent pain in the upper extremity (VAS>40)
* Patients with severe spasticity in the hand (MAS≥3)
* Patients with severe limitation of joint range of motion / contracture in the hand
* Patients who had fractures or operations in the upper extremity in the last 6 months
* Patients who received botulinum toxin injection to the upper extremity in the last 6 months
* Patients with skin ulcers
* Patients with severe visual impairment and severe depression
* Patients who cannot sit in a chair for more than 30 minutes
* Patients with a history of stroke or progressive neurodegenerative disease
* Patients with neuromuscular disease
* Patients with uncontrolled epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
American spinal cord injury association impairment scale | 15 minutes
  The ASIA Evaluation determines the level of injury in patients with spinal cord injury (SCI) based on the levels of sensory, motor, and neurologic injury. Neurological injury level (NLI): NLI refers to the most caudal segment of the spinal cord with normal sensory and antigravity motor function on both sides of the body, provided there is normal (integrated) sensory and motor function rostrally.
Sollerman hand function test | 60 minutes
  It consists of 20 different activities based on eight basic hand grips (pulp grip, lateral pinch, triple pinch, 5-finger pinch, diagonal volar grip, transverse volar grip, spherical volar grip, extension type grip). It also evaluates functional properties. Scoring of activities was done in the range of 0-4, according to the completion time of the activity. Failure to perform the activity 0, if it is performed in 60 seconds 1, if it is completed between 60-41 seconds or not with the desired grip pattern 2, if it is completed between 21-40 seconds and there is a minimum deviation in the grip pattern 3, if it is completed within 20 seconds with the specified grip pattern 4 points evaluated.The scoring rules were chosen so that subjects with normal hand function would achieve 80 points. As the score increases, the success rate of the test increases.
Nine Hole Peg Test | 20 minutes
  This test measures dexterity based on performance (in seconds). A wooden board with nine holes on it, 9 short wooden sticks and a box in which the wooden sticks can be placed are placed in front of the patient. Using the hand to be evaluated, the patient is asked to place the wooden sticks in the box into the holes on the panel as quickly as possible. Then, he is asked to put the sticks back into the box one by one. The completion time of the test is determined by a stopwatch. In this test, which evaluates manual dexterity based on performance, the success rate increases as the time gets shorter.
Box and block test | 30 minutes
  It is used to evaluate rough manual dexterity based on performance (time). 150 small wooden cubes are filled from the box with the patient's hand to be tested into the adjacent box. The patient is asked to throw one cube at a time into the semi-empty box. How many cubes are thrown in 60 seconds is counted. The result gives the score. How many cubes are thrown in 60 seconds is counted. The result gives the score. The higher the score, the higher the success rate.
Jamar pinchmeter | 5 minutes
  The hand grip strength of the participants will be measured with the 'Jamar Hand Dynamometer'. Measurements will be made with the shoulder adjacent to the trunk in adduction and neutral rotation, elbow 90 degrees flexed, wrist 0-30 degrees dorsiflexion and 0-15 degrees ulnar deviation with thumbs up. In the dominant and non-dominant hands, the measurements will be repeated three times (first right, then left and again right, etc.) with an interval of 5 seconds, and the average of the three measurements will be recorded in kilograms. The higher the score, the higher the success rate.
Jamar hand dynamometer | 5 minutes
  Finger grip strength will be evaluated with a 'Jamar digital pinchmeter'. Patients will be placed in a sitting position with the wrist in 90° flexion and the forearm in a neutral position. Measurements will be made bilaterally in three different positions as lateral, palmar and fingertip grips. Patients will be asked to squeeze with maximum force and each measurement will be made three times, and their averages will be recorded in kg.The higher the score, the higher the success rate

SECONDARY OUTCOMES:
Spinal cord injury independence scale | 15 minutes
  It is a test that determines the functional status in spinal cord injury. It is evaluated between 0-100 points. It consists of 17 items in total. This scale consists of self-care, respiratory-sphincter control and mobility subsections. : It is evaluated between 0-100 points. The higher the score, the higher the success rate.
Modified Ashworth Scale | 10 minutes
  In MAS, patients are evaluated over 5 points. 0; there is no increase in muscle tone, and 4 indicates that the extremity is rigid in the direction of flexion and extension.
Functional Independence Scale | 15 minutes
  It is a scale that evaluates the performance of individuals regarding activities of daily living. It consists of 18 items and evaluates the functions of individuals in 2 main sections: physical/motor function (13 items) and cognitive function (5 items). The items also include 6 subheadings (self-care, sphincter control,transfers, movement, communication, and social-perception).Each item is scored between 1-7; 1 indicates full assistance and 7 indicates complete independence. The total score ranges between 18-126 (fully dependent-fully independent).
Short form 36 | 15 minutes
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score was between 0 ( disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100 Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.Total score was between 0 ( disability) and 100 (no disability).

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA ADAR, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Sevda Adar, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No